CLINICAL TRIAL: NCT04387812
Title: Evaluation of the Frequency and Severity of Sleep Abnormalities in Patients With Parkinson's Disease (PD)
Brief Title: Evaluation of the Frequency and Severity of Sleep Abnormalities in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-20-NG-336-CTIL
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease; GBA Gene Mutation; Leucine-rich Repeat Kinase 2 (LRRK2) Gene Mutation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xtrodes home PSG system (Experimental): Wireless wearable system incorporates EEG, electrooculography (EOG) and EMG recordings over multiple nights in the home environment. The electrodes are printed on a thin sticker. These printed electrodes are marked by their conformity with the skin, light weight, ease of placement on the skin, and user comfort. The sleep-specific electrode array includes two surface EMG (electrodes 1 and 2), two EOG (electrodes 3 and 4) and four forehead EEG electrodes (electrodes 5-8) .
  Interventions: Device: Xtrodes home PSG system

INTERVENTIONS:
Device: Xtrodes home PSG system — Wireless, convenient and relies on actual recording of EMG, EOG and EEG in a home setting
  Other Names: Home PSG system

SUMMARY:
Sleep disturbances are one of the most common non-motor symptoms in PD, with an estimated prevalence as high as 40-90%. Sleep disturbances (particularly sleep duration, sleep fragmentation, Rapid Eye Movement (REM) sleep behavior disorder and sleep-disordered breathing) have been associated with an increased risk of neurodegeneration and are an independent risk for cognitive decline and dementia in PD.

Although much is currently unknown about sleep changes in PD, sleep-related symptoms are increasingly recognized as a major contributor to disease burden and reduced quality of life among people with PD. The "gold standard" evaluation of nocturnal sleep is polysomnographic monitoring (PSG).

This study proposes to use novel wireless skin electrodes and wearable sensors to provide a "home PSG test" incorporating several physiologic recordings, over multiple nights in the person's home, enabling the objective evaluation of night-to-night fluctuations.

DETAILED DESCRIPTION:
Background Sleep disturbances are one of the most common non-motor symptoms in PD, with an estimated prevalence as high as 40-90%. Sleep disturbances (particularly sleep duration, sleep fragmentation, Rapid Eye Movement (REM) sleep behaviour disorder and sleep-disordered breathing) have been associated with an increased risk of neurodegeneration and are an independent risk for cognitive decline and dementia in PD. The etiology of impaired sleep and alertness in PD is multifactorial and may be due to the interactions between internal and external factors such as primary sleep disorders, primary neurodegeneration, medication side effects, environmental conditions and genetic factors (either associated with sleep or associated with disease phenotype). Each can contribute to sleep disturbances alone or as modifiers, resulting in variability of presentation and symptoms, affecting both the diagnosis, and the treatment of these disorders. Although much is currently unknown about sleep changes in PD, sleep-related symptoms are increasingly recognized as a major contributor to disease burden and reduced quality of life among people with PD.

The "gold standard" evaluation of nocturnal sleep is polysomnographic monitoring (PSG). PSG consists of measuring neural function, eye movements, muscle activity, respiratory status and electrocardiography activity while the person sleeps over-night in a laboratory setting. This assessment allows for quantification of the different sleep stages during non-REM and REM, evaluation of their distribution over the course of the night, and the identification of impairments in each of these stages. However, PSG is time, cost and labor-intensive, may not reflect the typical behavior of the person due to the unfamiliar environment and irregular sleeping conditions, and more importantly, only provides information on one night of sleep.

In recent years, there is heightened interest in home-based sleep monitoring via wearable sensors to address these shortcomings. Body-fixed electrophysiological sensors can objectively quantify sleep quality, generating a detailed map of the person's sleeping pattern and nocturnal movements. They are relatively inexpensive enabling wide-spread use.

This study proposes to use novel wireless skin electrodes and wearable sensors to provide a "home PSG test" incorporating several physiologic recordings, over multiple nights in the person's home, enabling the objective evaluation of night-to-night fluctuations. By applying these novel tools to the study of people with PD as well as controls and subjects at risk for developing PD, the results of this study will open the door for using a new method for assessment of prodromal signs and disease progression.

Study objective

Main objective is to use the combined wearable system described above to evaluate sleep disturbances across a wide spectrum of PD disease severity: from the prodromal phase with individuals at risk to mild and advanced PD:

1. To investigate changes in sleep architecture and unique patterns of sleep in individuals at risk for developing PD (patients with confirmed RBD and carriers of mutations in the LRRK2 and GBA genes) that can help to better identify increased risk of disease.
2. To assess the frequency, severity and types of sleep disturbances in patients with PD across the disease spectrum.
3. To identify classifiers of sleep measures indicative of disease characteristics, severity and progression.
4. To assess the association between sleep disorders, disease severity, autonomic, motor, cognitive functions, and medication.

Subjects will be recruited and evaluated from the Laboratory for Early Markers of Neurodegeneration (LEMON) at the Neurological Institute at the Tel Aviv Medical Centre (TLVMC). All subjects will provide informed written consent as approved by each TLVMC's ethical committee and in accordance with the Helsinki agreement prior to participation.The 'Genetics in Parkinson's Study' registry will be used for initial recruitment of participants. This is a registry of participants (patients and family members who have undergone genetic testing in our lab previously and have agreed to allow contact for future studies (under Helsinki agreement of 05-069 and 07-0381). PD patients will be approached by their physician to provide consent to participate in the sleep study. Asymptomatic participants will be recruited from the registry or from public advertisements and word to mouth approach. Those willing to participate will be invited to LEMON for an assessment meeting. Subjects will be provided with a detailed explanation of the study protocol before being asked to sign the consent form.

Procedures:

After signing an informed written consent, participants will be asked about their current and medical history, sleep habits, dietary, alcohol and caffeine consumption and any medication they are receiving. Subjects will then undergo a through neurological assessment and blood pressure supine and standing, pulse rates, weight, height will be obtained.

A blood sample (15 cc) will be drawn to test the association to metabolic, hormonal and inflammatory mediators known to affect sleep (specifically: iron stores, thyroid function, and hemoglobin). Subjects will also undergo several performance based assessments and questionnaires on sleep and behavior.

All subjects will then be scheduled for a sleep polysomnography (PSG). Subjects will be invited to the sleep lab at TLVMC and asked to arrive at 9 pm and will be instructed on all procedures. Several body functions will be recorded during the PSG including brain activity, eye movement, oxygen and carbon dioxide blood levels, heart rate and rhythm, breathing rate and rhythm, the flow of air through the mouth and nose, body muscle movements, and chest and belly movement. The standard PSG will be fitted first and then the Xtrode system will be placed on the subject's face and the Axivity sensor will be placed on the subjects back (L4-5) using medical tape. This process should take approximately 45 minutes. After the systems are turned on, the subjects will be left in the quite room for a night sleep. The session will be video-taped to enable a comparison of movement with the wearable systems. The PSG and Xtrodes systems will be removed no later than 8 am the next morning.

Subjects will then be instructed on how to use the sleep "tattoo" at home. The system provided will include the controller, seven skin adhesives and a smartphone app, which will be used to obtain the data collected. Data is automatically transferred from the skin tattoo directly to the smartphone via a Bluetooth connection. The Axivity device which was placed on the lower back of the subjects will remain in place for the remaining 7 days. The device is waterproof thus there is no need for the subjects to don or doff the device until the end of the collection period. After the study, the systems will be returned to the medical centers for data transfer and analysis via carrier.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD (according to UK brain bank or Gelb criteria)
* Hohen and Yahr stages I-IV
* Age between 50-80
* First-degree healthy relatives, carriers of mutations in the LRRK2 and GBA genes
* Healthy volunteers
* Healthy subjects with confirmed RBD
* For patients with PD: only if they have a care partner at home who will be able to assist with the application of the technology
* Willing and able to sign an informed consent

Exclusion Criteria:

* Any neurological condition other than PD (e.g. Stroke, MSA, parkinsonism)
* Severe cognitive impairment (MoCA<24)
* Psychiatric disorders
* Low back pain or any orthopaedic problem or pain that will prevent the subject from sleeping in the sleep lab or wearing the wearable sensors
* For men: a beard (because of the tattoo adhesion

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in sleep architecture | From placing the system to disassembling, up to 1 week
  Frequency of RBD and severity of sleep interruptions

SECONDARY OUTCOMES:
MDS-UPDRS | Immediate after disassembling the system (day 7)
  MDS-UPDRS part III will be used to assess the relationship between sleep disorders and motor disability
REM Sleep Behavior Disorder Screening Questionnaire | Immediate after disassembling the system (day 7)
  Patient self-rating instrument assessing the subject's sleep behavior with short questions that have to be answered by either "yes" or "no".
The Non-Motor Scale | Immediate after disassembling the system (day 7)
  The Non-Motor Scale validated and commonly used 30-point questionnaire recognizes the non-motor difficulties often occur in PD. Areas covered include sleep, constipation, vision, smell, sexual problems and memory.
Geriatric Depression Scale | Immediate after disassembling the system (day 7)
  The Geriatric Depression Scale is a self report assessment used to identify depression in the elderly. The questionnaire consists of 15 yes/no questions; one point is assigned to each answer. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Anat Mirelman, PhD, Principal Investigator — Laboratory of Early Markers of Neurodegeneration (LEMON), TASMC
Locations (1):
- Tel Aviv Sourasky Medical Center, Neurology Department, Tel Aviv, Israel